CLINICAL TRIAL: NCT04972318
Title: Prospective, Randomized, Controlled Trial Assessing the Effects of a Driving-pressure Limiting STrAtegy for Patients With Acute Respiratory Distress Syndrome Due to coMmunIty-acquired pNeumoniA (STAMINA Trial)
Brief Title: Two Different Ventilatory Strategies in Acute Respiratory Distress Syndrome Due to Community-acquired Pneumonia
Acronym: STAMINA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate with no possibility to achieve pre specified sample size before funding ends.
Sponsor: Hospital do Coracao (Other)
Collaborators: Brazilian Research In Intensive Care Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: stamina_trial
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-06

CONDITIONS: Community-acquired Pneumonia; Acute Respiratory Distress Syndrome
Keywords: mechanical ventilation; positive end-expiratory pressure; community-acquired pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Respiratory Distress Syndrome | interventions — Physical Endurance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARDSNet strategy (Active Comparator): Patients will receive a mechanical ventilation strategy based on fixed values of positive end-expiratory pressure according to inspired fraction of oxygen.
  Plateau pressure will be limited at 30 cmH2O. This strategy will be mantained and monitored for 3 days, unless the patient dies or is extubated before.
  This arm is similar to the ARMA (Ventilation with Lower Tidal Volumes as Compared with Traditional Tidal Volumes for Acute Lung Injury and the Acute Respiratory Distress Syndrome) trial.
  Interventions: Procedure: ARDSNet ventilatory strategy
- STAMINA strategy (Experimental): Patients will receive a mechanical ventilation strategy based on positive end-expiratory pressure tailored to achieve the optimal respiratory system compliance and to have driving pressure limited to 14 cmH2O.
  Plateau pressure will be limited at 30 cmH2O. This strategy will be mantained and monitored for 3 days, unless the patient dies or is extubated before.
  Interventions: Procedure: Positive end-expiratory pressure titration with driving pressure control

INTERVENTIONS:
Procedure: Positive end-expiratory pressure titration with driving pressure control — Positive end-expiratory pressure will be tailored during a decremental maneuver (without a formal alveolar recruitment maneuver). The best positive end-expiratory pressure will be defined as the one associated with the higher respiratory system compliance, up to 20 cmH2O. Plateau pressure limit will be 30 cmH2O. If driving pressure remains elevated after optimal PEEP setting, tidal volume will be reduced to keep driving pressure below 14 cmH2O.
  Other Names: STAMINA
  Arms: STAMINA strategy
Procedure: ARDSNet ventilatory strategy — Positive end-expiratory pressure will be set according to fixed inspired oxygen fraction values.
  Arms: ARDSNet strategy

SUMMARY:
Randomized Controlled Trial Comparing Two Different Ventilatory Strategies in Acute Respiratory Distress Syndrome Due to Community-acquired Pneumonia. The control strategy will be based on ARDSNet approach. The intervention group will receive a different ventilatory strategy based on positive end-expiratory pressure tailored according to compliance and limited driving pressure.

DETAILED DESCRIPTION:
There is no consensus on the optimal ventilatory management of patients with community-acquired pneumonia that require mechanical ventilation and have acute respiratory distress syndrome. The traditional ventilatory approach (ARDSNet) is based on a fixed table for both end respiratory positive end-expiratory pressure according to inspired oxygen fraction. Alternatively, a strategy that tailors positive end-expiratory pressure according to compliance and limits driving pressure may be beneficial, but evidence is lacking.

We will perform an open label randomized controlled trial comparing both strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with community acquired pneumonia requiring invasive mechanical ventilation
* Bilateral pulmonary infiltrates on chest imaging not fully explained by fluid overload in the opinion of the attending physician
* One of the criteria below:
* Oxygen inspired fraction above 50% with a positive end-expiratory pressure of at least 8 cmH2O to main peripheral oxygen saturation above 93%, OR
* Arterial partial pressure of oxygen divided by inspired fraction of oxygen lower than 200 with PEEP values of at least 5 cmH2O

Exclusion Criteria:

* Patients with inclusion criteria for more than 36 hours
* Refusal of the patient´s legal representative
* Acute neurologic disease (stroke, brain trauma, or any disease that may cause intracranial hypertension)
* Patients with current airway fistula or barotrauma
* Patients on chronic home use of oxygen due to underlying lung disease
* Patients younger than 18 years
* Patients not on full code status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation free days | 28 days
  Number of days patient remains independent of mechanical ventilation

SECONDARY OUTCOMES:
Hospital Mortality | 90 days
  Whether the patient perished or not during hospitalization
Intensive Care Unit Mortality | 90 days
  Whether the patient perished or not during intensive care unit stay, truncated at 28 days
Need for rescue therapies for refractory hypoxemia | 28 days
  Need for extracorporeal membrane oxygenation, alveolar recruitment maneuver, or inhaled nitroux oxide, truncated at 28 days
Occurrence of barotrauma | 28 days
  Occurrence of either subcutaneous emphysema, pneumothorax or pneumatocele, truncated at 28 days

OTHER OUTCOMES:
Oxygenation parameters (oxygenation index and fraction of arterial pressure of oxygen over inspired oxygen fraction) | 3 days
  Measurements of oxygenation in the first 3 days after enrollment (ratio between arterial partial pressure of oxygen over inspired fraction of oxygen, and oxygenation index, defined by mean airway pressure multiplied by fraction of inspired oxygen over arterial partial pressure of oxygen.
Driving Pressure during mechanical ventilation | 3 days
  Driving pressured, measured once daily and defined by airway plateau pressure minus positive end-expiratory pressure
Intensive Care Unit Free Days | 28 days
  Number of days the patient spend alive and out of the intensive care unit
Ventilatory Rate | 3 days
  Ventilatory Rate, measured daily, defined as minute ventilation (in liters) multiplied by arterial partial pressure of oxygen, divided by 37.5 multiplied by patient weight (in kilograms) multiplied by 100

CONTACTS AND LOCATIONS:
Overall Officials: Israel S Maia, MSc, Study Chair — HCor Research Institute; Bruno Tomazini, MD, Principal Investigator — HCor Research Institute
Locations (6):
- Brazil (6):
  - Associação Evangélica Beneficente de Londrina - Hospital Evangélico de Londrina, Londrina, Paraná
  - Hospital São José, Criciúma, Santa Catarina
  - Hospital Nereu Ramos, Florianópolis, Santa Catarina
  - Centro Hospitalar Unimed, Joinville, Santa Catarina
  - Hospital do Coracao, São Paulo
  - BP-A Beneficiência Portuguesa de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after publication of primary results
Access Criteria: Submission of a statistical analysis plan for the purposed analyses. Compliance with Brazilian. data privacy law.

REFERENCES:
- [Derived] Maia IS, Cavalcanti AB, Tramujas L, Veiga VC, Oliveira JS, Sady ERR, Barbante LG, Nicola ML, Gurgel RM, Damiani LP, Negrelli KL, Miranda TA, Laranjeira LN, Tomazzini B, Zandonai C, Pincelli MP, Westphal GA, Fernandes RP, Figueiredo R, Sartori Bustamante CL, Norbin LF, Boschi E, Lessa R, Romano MP, Miura MC, Soares de Alencar Filho M, Ces de Souza Dantas V, Barreto PA, Hernandes ME, Grion C, Laranjeira AS, Mezzaroba AL, Bahl M, Starke AC, Biondi R, Dal-Pizzol F, Caser E, Thompson MM, Padial AA, Leite RT, Araujo G, Guimaraes M, Aquino P, Lacerda F, Hoffmann Filho CR, Melro L, Pacheco E, Ospina-Tascon G, Ferreira JC, Calado Freires FJ, Machado FR, Zampieri FG; BRICNet. Effect of a driving pressure-limiting strategy for patients with acute respiratory distress syndrome secondary to community-acquired pneumonia: the STAMINA randomised clinical trial. Br J Anaesth. 2025 Mar;134(3):693-702. doi: 10.1016/j.bja.2024.10.012. Epub 2024 Nov 26. PMID 39592365